CLINICAL TRIAL: NCT04388592
Title: MS Wellness Navigator: The Effect of Nurse Practitioner (NP-led) Care on Mood, Anxiety and Health Related Quality of Life in People With Multiple Sclerosis - A Randomized Trial
Brief Title: The Effect of Nurse Practitioner (NP-led) Care Upon Mood in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University Hospital Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00069595
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-06

CONDITIONS: Multiple Sclerosis; Nurse's Role
Keywords: multiple sclerosis; nurse's role; depression and anxiety; quality of life; patient satisfaction
MeSH Terms: conditions — Multiple Sclerosis; Depression; Anxiety Disorders; Patient Satisfaction | interventions — Nurse Practitioners

STUDY DESIGN:
Intervention Model Description: A parallel prospective randomized controlled trial with two equal groups, testing for superiority, with the patient as the unit of randomization.
Who Masked: Outcomes Assessor
Masking Description: The research team will randomize consented patients who meet inclusion criteria on a 1:1 ratio on a centralized secure website. Block randomization (using variable block sizes) will be used to ensure there are equal participants in the intervention and control arms and to further conceal allocation. Participants will be randomized to either the intervention group of NP-led care or the control group of standard care provided by community neurologist and registered nurse. Due to the nature of the intervention, blinding of the providers or patients will not be possible. However, the statistician will be blinded as to which group represents the intervention and control. All participants will be given appointment with the NP, either within 4 to 6 weeks if randomized to the intervention arm, or at 6 months after study conclusion if in usual care arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse practitioner (NP)-led care arm (Experimental): The patient randomized to the NP intervention arm will be contacted by the NP to be scheduled for an NP appointment within 4 to 6 weeks from the date of the referral. The NP consultation will include patient history, physical examination, symptomatic management strategies as appropriate (eg: bladder and bowel management strategies, fatigue management, depression, anxiety, spasticity etc), discussion of mental and physical health resources for symptomatic treatment, support, physical and mental health resources to optimize functioning (eg: home care, physical/occupational therapy referral) and quality of life. There will be NP followup, in person or by phone or videoconferencing at 3 months, and 6 months. The NP will be using the electronic medical record offered by Alberta Health Services.
  Interventions: Other: Nurse Practitioner (NP) Led Care Arm
- Usual Care Arm (No Intervention): Those patients randomized to the usual care arm (community neurologist and registered nurses) will be contacted by the NP to be scheduled for an NP appointment in 6 months, so that every participant is given the opportunity to meet with the NP, after their involvement in the study has concluded. During the six-month period, patients randomized to the control group will receive usual care from community neurologists and MS registered nurses or family physicians. The care will be delivered according to standard practices, and follow-up visits will be conducted according to the various neurologists' or family physicians' practices.

INTERVENTIONS:
Other: Nurse Practitioner (NP) Led Care Arm — The NP will conduct baseline consultation visits with the participants and their caregivers (if applicable). They will then initiate treatment for the participant's symptoms as appropriate (ie: depression treatment for depressive symptoms, fatigue management strategies), connect to resources in the community as needed (ie: rehabilitation programs, home care support, psychologist support) to optimize functioning. There will be scheduled follow visits and/or phone calls with the NP at 3 and 6 months.
  Arms: Nurse practitioner (NP)-led care arm

SUMMARY:
MS is the leading cause of non-traumatic disability in young adults. Canada and Alberta, have the highest prevalence of people with multiple sclerosis (PwMS) in the world. To keep PwMS as functional as possible, a multi-disciplinary team is considered essential in the approach to treating people with MS. Because of the high numbers of PwMS in Northern Alberta, private-practice general neurologists provide care to a large number of PwMS outside of a multi-disciplinary tertiary care setting. It is challenging for these general neurologists with busy office practices to deliver optimal care to PwMS who have high care needs. The investigators wish to evaluate the effects of nurse practitioner (NP) led care for PwMS on their depression and anxiety levels at 3 and 6 months compared to "usual care' (community neurologists and MS registered nurses) in addition to measuring quality of life for PwMS and their caregivers, fatigue levels, monitor their outpatient healthcare usage and patient's satisfaction of care provided. The investigators wish to conduct a prospective randomized controlled trial examining NP intervention care for PwMS. It is hypothesized that PwMS whose care is managed by an NP will have less depression and anxiety (as measured by the Hospital Anxiety and Depression Scale - HADS) at 3 months.

DETAILED DESCRIPTION:
Background:

MS is the leading cause of non-traumatic disability in young adults. It is most commonly diagnosed in people between the ages of 20 to 50, causing visible and invisible disability that limits functioning and progresses over time. Canada has one of the highest prevalence of MS in the world; Alberta has the highest rate of MS in Canada (340/100 000 population). Having MS is associated with significant economic, physical and psychological burdens on the individual with corresponding burden upon society.

Global approach to treating and supporting PwMS has become multidisciplinary, multi-pronged and increasingly complex; MS impacts a person's physical, psychological and social well-being. Despite advances in healthcare for PwMS in the 21st century, multiple studies have reported a number of unmet care needs for PwMS: in areas of healthcare delivery, education, counselling and psychological support, and in supporting their informal caregivers. Recently, a study of over 1000 PwMS, reported that a higher number of reported health and social care-related unmet needs predicted lower health related quality of life, with all domains of the EQ5D-3L as being important.

PwMS prefer multidisciplinary care, recommended as essential by international multiple sclerosis experts. It has been reported that NPs are well-placed providers for PwMS, with their expertise in chronic disease management and quality of life approach. A recent integrative review identified three themes to the role of the MS nurse specialist: (1) longitudinal care co-coordinator; (2) care provider; and (3) expert resource. In one questionnaire study, PwMS indicated that they preferred contacting the specialized MS nurse above other health professionals. In addition, having NPs to enhance the multi-disciplinary team could potentially provide healthcare cost-savings: in the United States, NP-led care was reported to be cost-saving in comparison to physician-led care.

Private-practice general neurologists and family doctors provide care to approximately 2000 PwMS outside of a tertiary multi-disciplinary clinic setting with a wide catchment area extending across Central and Northern Alberta, Northern BC, Saskatchewan and Northwest Territories. It is challenging for general neurologists and family doctors to balance care of PwMS with the pressures of busy office practices in a fee-for-service setting.

There have been few controlled randomized trials comparing NP-led care vs usual care for people with chronic diseases. One demonstrated clear benefits of NP involvement in managing people with chronic pain, reporting better pain control, coping, and use of pain medication by those followed by an NP, while another trial reported better outcomes for people with Parkinson's disease randomized to multidisciplinary team care with an NP vs care by a general neurologist. The investigators wish to follow a similar protocol to Smigorowsky et al, who studied the impact of NP-led care for people with atrial fibrillation.

The study's aim is to evaluate the effects of NP-led care for PwMS on their depression and anxiety levels at 3 months and 6 months compared to 'usual care' (community neurologists' care and MS registered nurses), in addition to measuring quality of life for PwMS and their caregivers, fatigue levels, outpatient healthcare visits and phone calls, and to measure patients' satisfaction of the care provided.

Design: The investigators will conduct a prospective randomized controlled trial with two equal groups. It is hypothesized that PwMS whose care is managed by an NP would have less depression and anxiety (as measured by the Hospital Anxiety and Depression Scale - HADS) at 3 months.

The randomized controlled trial will be conducted in a distributed, outreach model, in the offices of seven community neurologists who follow PwMS as a part of their general neurology private practices. Family doctors will be able to refer patients with MS directly to the NP, if not followed by any neurologist, through the MS clinic referral process already established. The research team will randomize consented participants who meet inclusion criteria on a 1:1 ratio on a centralized secure website.

Participants will be randomized to NP intervention of providing care for 6 months vs usual care provided by their regular neurologist, a MS registered nurse or their family doctors.

3.10 Primary and Secondary Outcomes: The primary outcome will be the difference in change in HADS-D and HADS-A scores between intervention and control groups at 3 months. Secondary outcomes will include difference in change in: (a) HADS-D and HADS-A scores at 6 months; (b) Euro Quality of Life 5D (EQ5D) at 3 and 6 months; (c) Modified Fatigue Impact Scale (MFIS) score at 3 and 6 months; CAREQOL-MS - caregiver health-related quality of life in MS questionnaire for those participant caregivers, who agree to participate in a questionnaire at baseline, 3 months and 6 months, and number of healthcare outpatient visits/interactions during the study period.

Participants' satisfaction with the level of care provided to them will be measured at 6 months using a validated Consultant Satisfaction Questionnaire (CSQ).

3.11 Recruitment, consent and data collection: Recruitment will be done through a few methods, due to potential participants being recruited from various community neurologists' offices and family doctors' practices in Northern Alberta: (1)There are seven community neurologists who will participate in recruitment through their practices. (2) PwMS who are followed primarily by a family physician will be referred by their family physicians directly to the NP via the tertiary MS Clinic fax (3) Caregivers will be approached through the PwMS, if the PwMS consents to participating in the study. After informed consent, PwMS and their informal caregivers (where applicable) will be invited to complete the questionnaires (HADS-D/HADS-A, EQ5D, MSIF, CAREQOL-MS at baseline, 3 months and 6 months with a participant diary of outpatient visits and phone calls with healthcare providers submitted at 3 and 6 months, and a consultant satisfaction questionnaire completed at 6 months. The questionnaires will take around 10 to 15 minutes each time to complete.

3.12 Sample Size: Using the information from Honarmand and Feinstein [Baseline scores and standard deviation (SD)], and the following assumptions 90% power and a two-sided alpha of 0.05, a total sample size of 200 (100 in each group) will be required to detect 1.5 difference between the intervention and the control groups.

3.14 Statistical Analyses: Data analysis will be performed. Categorical variables will be reported using frequency and percentage and continuous variables will be reported using mean (SD) or median [Interquartile range (IQR)] as appropriate. Univariable analysis will be conducted to determine if there was a statistical significance between the outcomes from baseline to three months and six months, respectively. All test assumptions will be checked during the data analysis process. Independent T-test will be used to assess the primary (HADS-D and HADS-A at 3 months) and secondary outcomes (HADS-D and HADS-A at 6 months, EQ5D, and MFIS). The consultant satisfaction survey will be analyzed as continuous variables, with the overall satisfaction score being calculated as a sum of the scales of each question.

3.15 Validity and Reliability: The questionnaires used in the study have been tested for validity and reliability in studies involving PwMS. Three papers report total HADS scores in PwMS.The EQ5D quality of life measure is commonly used in the MS population, and the MSIF is a standard measurement of fatigue in MS, as has the CAREQOL-MS, a caregiver quality of life survey for those caring for PwMS. Satisfaction with healthcare provider care will be measured by the overall mean score of the consultation satisfaction questionnaire (CSQ) completed at the 6 month follow-up visit. The CSQ is a self-administered tool with 18 questions using a 5-point Likert scale, ranging from strongly agree to strongly disagree. It measures 3 factors of the healthcare provider interaction: (1) professional aspects; (2) depth of patient relationship with provider; and (3) perceived length of consultation. Higher scores indicate higher satisfaction. We will reduce biases through using objective measures to examine the effects of NP-led care intervention. It is impossible to blind the participants for the intervention. It is important that all participants are offered NP intervention to minimize bias from those in either the intervention or control arm, by having those participants randomized to the control arm being seen by the NP at 6 months, after their involvement in the study has concluded. That way, all participants in the study are offered appointment with the NP, either within 4 weeks for the intervention arm vs at 6 months for the control arm.

3.16 Ethical considerations: The research protocol was reviewed and approved by the Health Research Ethics Board of the University of Alberta.(approval number Pro00069595) PwMS will be able to be referred to the NP by community neurologists and family doctors outside of participating in the study, if they decline to participate in the study.

3.17 Conclusion: To the investigators' knowledge, there have been no studies examining effects of NP-intervention of care for PwMS in a prospective, randomized and controlled clinical trial. Findings of this study will contribute to ways in which the multi-disciplinary care for PwMS and their caregivers could be enhanced by the addition of a specialized NP to aid general community neurologist practices in care delivery to PwMS outside of tertiary MS clinic settings. This study will evaluate the effects of nurse practitioner intervention depression and anxiety levels in PwMS and their informal caregivers. The evidence gained from this study will provide information on how nurse practitioners enhance the care and potentially resolve identified unmet needs for PwMS when introduced as part of a multi-disciplinary team approach for general neurologists working in a distributed community setting.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years of age
* a MS diagnosis (by 2010 MacDonald MS criteria (Polman et al 2011)
* Followed by a private-practice general neurologist and/or family doctor in the Northern Alberta region
* Willingness to give consent
* Ability to complete questionnaires
* Willingness to attend outpatient visits with NP
* English-speaking
* Were able to use a computer
* Initially, we limited inclusion to those who are experiencing disability from their MS (Expanded Disability status Scale (EDSS) 3.0 to 8.5 . In 2018, due to poor recruitment, the inclusion criteria were opened to include any PwMS and was not limited to disability level.

Exclusion Criteria:

* Under the age of 18 years old
* Unable to provide consent
* Unable to attend appointments with the NP
* Did not speak English
* Referred to or followed by neurologists within the tertiary University MS clinic setting
* Those who had central nervous system inflammatory disorders other than MS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants are enrolled as how they report themselves to be.
Enrollment: 248 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Difference in Change in Hospital Anxiety & Depression Scale - Depression (HADS-D) and Hospital Anxiety & Depression Scale-Anxiety (HADS-A) scores | 3 months
  Hospital Anxiety & Depression Scale (D subcategory for depression levels, A subcategory for anxiety levels). This is a common depression and anxiety measurement instrument used in multiple sclerosis. Minimum score is 0, and maximum score is 21. Higher scores indicate worse outcome.
  Three papers report total HADS scores in PwMS. Using the information from Honarmand and Feinstein [Baseline scores and standard deviation (SD)] and the following assumptions 90% power and a two-sided alpha of 0.05, a total sample size of 200 (100 in each group) was required to detect 1.5 difference between the intervention and the control groups. This sample size was inflated to 220 to account for possible dropouts, losses to follow-up and withdrawals of consent.

SECONDARY OUTCOMES:
Difference in Change in Hospital Anxiety & Depression Scale - Depression (HADS-D) and Hospital Anxiety & Depression Scale-Anxiety (HADS-A) scores | 6 months
  Hospital Anxiety & Depression Scale (D subcategory for depression levels, A subcategory for anxiety levels). This is a common depression and anxiety measurement instrument used in multiple sclerosis. Minimum score is 0, and maximum score is 21. Higher scores indicate worse outcome.
  Three papers report total HADS scores in PwMS. Using the information from Honarmand and Feinstein [Baseline scores and standard deviation (SD)] and the following assumptions 90% power and a two-sided alpha of 0.05, a total sample size of 200 (100 in each group) was required to detect 1.5 difference between the intervention and the control groups. This sample size was inflated to 220 to account for possible dropouts, losses to follow-up and withdrawals of consent.
Difference in Change in Euro Quality of Life Measurement (EQ5D) | 3 and 6 months
  The EQ5D quality of life measure is used in the MS population (Kuspinar & Mayo, 2014), and is the main quality of life measure preferred by Alberta Health Services. There is a descriptive element to the EQ5D that represents values around the level of reported problems in each of the 5 domains, with higher scores being worse. The 5 domains are around (1) mobility; (2) self-care; (3) usual activities; (4) pain/discomfort; and (5) anxiety/depression. The index is calculated by deducting the appropriate weights from 1 and comparing to population norms in a value set.
Difference in Change Modified Fatigue Impact Scale (MFIS) score | 3 and 6 months
  Fatigue is one of the most common symptoms for people with MS. The MSIF is a standard, validated measurement of fatigue in MS. The MFIS is a self-report instrument in which participants are asked to rate how often fatigue has affected them in the previous 4 weeks in relation to statements (0 = never to 4 = almost always). Items on the MFIS can be aggregated into subscales (physical, cognitive and psychosocial) as well as into a total MFIS score. The total MFIS score can be a minimum of 0 to 84, computed by adding the scores on the physical, cognitive and psychosocial subscales.
Qualitative Consultant Satisfaction Questionnaire (CSQ) | 6 months
  Participants' satisfaction with the level of care provided to them will be measured at 6 months using the validated Consultant Satisfaction Questionnaire (CSQ). CSQ consists of 18 Likert scale questions, ranging from 1= strongly disagree to 5 = strongly agree, with the higher score indicating higher patient satisfaction. Satisfaction with healthcare provider care will be measured by the overall mean score of the consultation satisfaction questionnaire (CSQ) completed at the 6 month follow-up visit. The CSQ is a self-administered tool with 18 questions using a 5-point Likert scale, ranging from strongly agree to strongly disagree. It measures 3 factors of the healthcare provider interaction: (1) professional aspects; (2) depth of patient relationship with provider; and (3) perceived length of consultation. Higher scores indicate higher satisfaction.
Difference in Change in Caregiver Health-Related Quality of Life in MS (CAREQOL-MS) | 3 and 6 months
  CAREQOL-MS measures caregiver health-related quality of life (HRQOL) in multiple sclerosis (MS) (CAREQOL-MS) The CAREQOL-MS consists of 24 items using a 5 point Likert-type scale (higher scores reflecting worse health related quality of life). Dimensions of the CAREQOL-MS include subscale I (physical burden and global health - 8 items); subscale II (social impact - 5 items); subscale III (emotional impact - 6 items); subscale IV (need of help - 3 items); and subscale V (emotional reactions - 2 items). Minimum total score is 24 and maximum total score is 120.
Number of Participant Outpatient Healthcare Interactions/Visits | 3 and 6 months
  Participants will keep a participant diary, outlining number of outpatient visits and phone calls to their neurologists, family physicians, registered nurses, pharmacists, physiotherapists, occupational therapists and other allied health professionals (such as massage therapists, chiropractors, dieticians etc). Higher numbers of recorded visits on the diary correspond to a greater number of outpatient healthcare visits and interactions. Minimum score is 0, and there is no upper limit score.

CONTACTS AND LOCATIONS:
Overall Officials: Penelope Smyth, MD, FRCPC, Principal Investigator — University of Alberta; Ross Tsuyuki, PharmD, MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amankwah N, Marrie RA, Bancej C, Garner R, Manuel DG, Wall R, Fines P, Bernier J, Tu K, Reimer K. Multiple sclerosis in Canada 2011 to 2031: results of a microsimulation modelling study of epidemiological and economic impacts. Health Promot Chronic Dis Prev Can. 2017 Feb;37(2):37-48. doi: 10.24095/hpcdp.37.2.02. PMID 28273039
- [Background] Atlas of MS 2013: mapping MS around the world. (2013). Retrieved May 6, 2020, from https://www.msif.org/wp-content/uploads/2014/09/Atlas-of-MS.pdf
- [Background] Baker R. Development of a questionnaire to assess patients' satisfaction with consultations in general practice. Br J Gen Pract. 1990 Dec;40(341):487-90. PMID 2282225
- [Background] Benito-Leon J, Rivera-Navarro J, Guerrero AL, de Las Heras V, Balseiro J, Rodriguez E, Bello M, Martinez-Martin P; caregiver quality of life in multiple sclerosis (CAREQOL-MS) Study Group. The CAREQOL-MS was a useful instrument to measure caregiver quality of life in multiple sclerosis. J Clin Epidemiol. 2011 Jun;64(6):675-86. doi: 10.1016/j.jclinepi.2010.08.003. Epub 2010 Nov 11. PMID 21071173
- [Background] Borreani C, Bianchi E, Pietrolongo E, Rossi I, Cilia S, Giuntoli M, Giordano A, Confalonieri P, Lugaresi A, Patti F, Grasso MG, de Carvalho LL, Palmisano L, Zaratin P, Battaglia MA, Solari A; PeNSAMI project. Unmet needs of people with severe multiple sclerosis and their carers: qualitative findings for a home-based intervention. PLoS One. 2014 Oct 6;9(10):e109679. doi: 10.1371/journal.pone.0109679. eCollection 2014. PMID 25286321
- [Background] Broderick JE, Keefe FJ, Bruckenthal P, Junghaenel DU, Schneider S, Schwartz JE, Kaell AT, Caldwell DS, McKee D, Reed S, Gould E. Nurse practitioners can effectively deliver pain coping skills training to osteoarthritis patients with chronic pain: A randomized, controlled trial. Pain. 2014 Sep;155(9):1743-1754. doi: 10.1016/j.pain.2014.05.024. Epub 2014 May 24. PMID 24865795
- [Background] Buchanan RJ, Radin D, Huang C. Caregiver burden among informal caregivers assisting people with multiple sclerosis. Int J MS Care. 2011 Summer;13(2):76-83. doi: 10.7224/1537-2073-13.2.76. PMID 24453708
- [Background] Buerhaus, P. (2018). Nurse Practitioners: a solution to America's primary care crisis: American Enterprise Institute.
- [Background] GBD 2016 Neurology Collaborators. Global, regional, and national burden of neurological disorders, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):459-480. doi: 10.1016/S1474-4422(18)30499-X. Epub 2019 Mar 14. PMID 30879893
- [Background] Fiest KM, Walker JR, Bernstein CN, Graff LA, Zarychanski R, Abou-Setta AM, Patten SB, Sareen J, Bolton JM, Marriott JJ, Fisk JD, Singer A, Marrie RA; CIHR Team Defining the Burden and Managing the Effects of Psychiatric Comorbidity in Chronic Immunoinflammatory Disease. Systematic review and meta-analysis of interventions for depression and anxiety in persons with multiple sclerosis. Mult Scler Relat Disord. 2016 Jan;5:12-26. doi: 10.1016/j.msard.2015.10.004. Epub 2015 Oct 19. PMID 26856938
- [Background] Fisk JD, Pontefract A, Ritvo PG, Archibald CJ, Murray TJ. The impact of fatigue on patients with multiple sclerosis. Can J Neurol Sci. 1994 Feb;21(1):9-14. PMID 8180914
- [Background] Forbes A, While A, Mathes L, Griffiths P. Health problems and health-related quality of life in people with multiple sclerosis. Clin Rehabil. 2006 Jan;20(1):67-78. doi: 10.1191/0269215506cr880oa. PMID 16502752
- [Background] Giovannoni G, Butzkueven H, Dhib-Jalbut S, Hobart J, Kobelt G, Pepper G, Sormani MP, Thalheim C, Traboulsee A, Vollmer T. Brain health: time matters in multiple sclerosis. Mult Scler Relat Disord. 2016 Sep;9 Suppl 1:S5-S48. doi: 10.1016/j.msard.2016.07.003. Epub 2016 Jul 7. PMID 27640924
- [Background] Hobart J, Bowen A, Pepper G, Crofts H, Eberhard L, Berger T, Boyko A, Boz C, Butzkueven H, Celius EG, Drulovic J, Flores J, Horakova D, Lebrun-Frenay C, Marrie RA, Overell J, Piehl F, Rasmussen PV, Sa MJ, Sirbu CA, Skromne E, Torkildsen O, van Pesch V, Vollmer T, Zakaria M, Ziemssen T, Giovannoni G. International consensus on quality standards for brain health-focused care in multiple sclerosis. Mult Scler. 2019 Nov;25(13):1809-1818. doi: 10.1177/1352458518809326. Epub 2018 Nov 1. PMID 30381987
- [Background] Holland NJ, Schneider DM, Rapp R, Kalb RC. Meeting the needs of people with primary progressive multiple sclerosis, their families, and the health-care community. Int J MS Care. 2011 Summer;13(2):65-74. doi: 10.7224/1537-2073-13.2.65. PMID 24453707
- [Background] Honarmand K, Feinstein A. Validation of the Hospital Anxiety and Depression Scale for use with multiple sclerosis patients. Mult Scler. 2009 Dec;15(12):1518-24. doi: 10.1177/1352458509347150. Epub 2009 Nov 13. PMID 19965520
- [Background] Jones KH, Ford DV, Jones PA, John A, Middleton RM, Lockhart-Jones H, Osborne LA, Noble JG. A large-scale study of anxiety and depression in people with Multiple Sclerosis: a survey via the web portal of the UK MS Register. PLoS One. 2012;7(7):e41910. doi: 10.1371/journal.pone.0041910. Epub 2012 Jul 30. PMID 22860028
- [Background] Kuspinar A, Mayo NE. A review of the psychometric properties of generic utility measures in multiple sclerosis. Pharmacoeconomics. 2014 Aug;32(8):759-73. doi: 10.1007/s40273-014-0167-5. PMID 24846760
- [Background] Lonergan R, Kinsella K, Fitzpatrick P, Duggan M, Jordan S, Bradley D, Hutchinson M, Tubridy N. Unmet needs of multiple sclerosis patients in the community. Mult Scler Relat Disord. 2015 Mar;4(2):144-50. doi: 10.1016/j.msard.2015.01.003. Epub 2015 Feb 3. PMID 25787190
- [Background] Maloni H, Hillman L. Multidisciplinary Management of a Patient With Multiple Sclerosis: Part 2. Nurses' Perspective. Fed Pract. 2015 Apr;32(Suppl 3):17S-19S. No abstract available. PMID 30766114
- [Background] McCabe MP, Ebacioni KJ, Simmons R, McDonald E, Melton L. Unmet education, psychological and peer support needs of people with multiple sclerosis. J Psychosom Res. 2015 Jan;78(1):82-7. doi: 10.1016/j.jpsychores.2014.05.010. Epub 2014 Jun 5. PMID 25516288
- [Background] Meehan M, Doody O. The role of the clinical nurse specialist multiple sclerosis, the patients' and families' and carers' perspective: An integrative review. Mult Scler Relat Disord. 2020 Apr;39:101918. doi: 10.1016/j.msard.2019.101918. Epub 2020 Jan 3. PMID 31927154
- [Background] Montanari E, Rottoli M, Maimone D, Confalonieri P, Plewnia K, Frigo M, Francia A, Pala A, Losignore NA, Ragonese P, Veneziano A; POSIDONIA study group. A 12-month prospective, observational study evaluating the impact of disease-modifying treatment on emotional burden in recently-diagnosed multiple sclerosis patients: The POSIDONIA study. J Neurol Sci. 2016 May 15;364:105-9. doi: 10.1016/j.jns.2016.02.047. Epub 2016 Feb 20. PMID 27084226
- [Background] Nourbakhsh B, Julian L, Waubant E. Fatigue and depression predict quality of life in patients with early multiple sclerosis: a longitudinal study. Eur J Neurol. 2016 Sep;23(9):1482-6. doi: 10.1111/ene.13102. Epub 2016 Jul 14. PMID 27416110
- [Background] Patti F, Amato MP, Battaglia MA, Pitaro M, Russo P, Solaro C, Trojano M. Caregiver quality of life in multiple sclerosis: a multicentre Italian study. Mult Scler. 2007 Apr;13(3):412-9. doi: 10.1177/1352458506070707. Epub 2007 Jan 29. PMID 17439911
- [Background] Ponzio M, Tacchino A, Vaccaro C, Traversa S, Brichetto G, Battaglia MA, Uccelli MM. Unmet needs influence health-related quality of life in people with multiple sclerosis. Mult Scler Relat Disord. 2020 Feb;38:101877. doi: 10.1016/j.msard.2019.101877. Epub 2019 Nov 29. PMID 31812039
- [Background] Puhan MA, Frey M, Buchi S, Schunemann HJ. The minimal important difference of the hospital anxiety and depression scale in patients with chronic obstructive pulmonary disease. Health Qual Life Outcomes. 2008 Jul 2;6:46. doi: 10.1186/1477-7525-6-46. PMID 18597689
- [Background] Puhan MA, Gaspoz JM, Bridevaux PO, Schindler C, Ackermann-Liebrich U, Rochat T, Gerbase MW. Comparing a disease-specific and a generic health-related quality of life instrument in subjects with asthma from the general population. Health Qual Life Outcomes. 2008 Feb 15;6:15. doi: 10.1186/1477-7525-6-15. PMID 18279510
- [Background] Smigorowsky MJ, Norris CM, McMurtry MS, Tsuyuki RT. Measuring the effect of nurse practitioner (NP)-led care on health-related quality of life in adult patients with atrial fibrillation: study protocol for a randomized controlled trial. Trials. 2017 Aug 3;18(1):364. doi: 10.1186/s13063-017-2111-4. PMID 28774317
- [Background] van der Marck MA, Bloem BR, Borm GF, Overeem S, Munneke M, Guttman M. Effectiveness of multidisciplinary care for Parkinson's disease: a randomized, controlled trial. Mov Disord. 2013 May;28(5):605-11. doi: 10.1002/mds.25194. Epub 2012 Nov 19. PMID 23165981
- [Background] The way forward: Alberta's multiple sclerosis partnership. (2013). Retrieved May 6, 2020, from https://open.alberta.ca/publications/9781460108574
- [Background] Ward-Abel, N., Mutch, K., & Huseyin, H. (2013). Demonstrating that multiple sclerosis specialist nurses make a difference to patient care (Vol. 6): British Journal of Neuroscience Nursing.
- [Derived] Smyth P, Watson KE, Al Hamarneh YN, Tsuyuki RT. The effect of nurse practitioner (NP-led) care on health-related quality of life in people with multiple sclerosis - a randomized trial. BMC Neurol. 2022 Jul 25;22(1):275. doi: 10.1186/s12883-022-02809-9. PMID 35879701